CLINICAL TRIAL: NCT04114019
Title: The Effect of Pelvic Floor Physiotherapy on Vaginal Elasticity as Measured by a Vaginal Tactile Imager
Brief Title: The Effect of Pelvic Floor Physiotherapy on Vaginal Elasticity
Status: Withdrawn | Type: Observational
Why Stopped: The study device became unavailable for use.
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Principal Investigator, Rambam Health Care Campus
Other Study IDs: 0327-19-RMB
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stress urinary incontinence: Women suffering from stress urinary incontinence
  Interventions: Diagnostic Test: Vaginal tactile imager

INTERVENTIONS:
Diagnostic Test: Vaginal tactile imager — Vaginal elasticity evaluation using a vaginal tactile imager

SUMMARY:
Women suffering from stress urinary incontinence are offered pelvic floor physiotherapy as an optional treatment. Strengthening of the pelvic floor is measured to date by manual examination and lacks precise evaluation. The vaginal tactile imager assists in evaluation of the changes in the pelvic floor after physiotherapy.

DETAILED DESCRIPTION:
Women with stress urinary incontinence will undergo 6-10 pelvic floor strengthening physiotherapy sessions. The participants will undergo a short examination of vaginal elasticity using a vaginal tactile imager prior to beginning physiotherapy and additional examinations after 6 treatments, 10 treatments and 3 and 6 months post-treatment cessation.

ELIGIBILITY:
Inclusion Criteria:

* women suffering from stress urinary incontinence.

Exclusion Criteria:

* women suffering from urge urinary incontinence.
* women suffering of mixed urinary incontinence.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Women between 18-70 years of age, suffering from stress urinary incontinence, referred to pelvic floor physiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Vaginal Elasticity | From the treatment cessation up to 6 months post-treatment
  Changes in vaginal elasticity post physiotherapy

SECONDARY OUTCOMES:
Stress urinary incontinence | From the treatment cessation up to 6 months post-treatment
  Improvement in the urogenital distress inventory questionnaire score (range 0-15)

CONTACTS AND LOCATIONS:
Overall Officials: Roy Lauterbach, MD, Principal Investigator — Rambam Health Care Campus

IPD SHARING:
Plan to Share IPD: No